CLINICAL TRIAL: NCT04037319
Title: Atrial Fibrillation After Resection (AFAR): A PROGRESS III Study
Brief Title: Atrial Fibrillation After Surgery for Colorectal Cancer
Acronym: AFAR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: STH20223
Record Dates: First submitted 2019-06-26; First posted 2019-07-30 (Actual); Last update posted 2021-10-08 (Actual); Status verified 2021-01

CONDITIONS: Colorectal Cancer; Atrial Fibrillation New Onset
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Electrocardiography, Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Main cohort: Will undergo surgery for colorectal cancer with curative intent as planned by local cancer multidisciplinary team.
  Interventions: Diagnostic Test: 24 Hour Holter Monitor

INTERVENTIONS:
Diagnostic Test: 24 Hour Holter Monitor — 24 hour holter monitor to be performed pre-operatively, and at day 30 and 90 post-operatively.

SUMMARY:
This study will report the incidence of atrial fibrillation after elective colorectal cancer resection in the over 65 age group. This will be used to validate a risk model for the development of post-operative atrial fibrillation.

Eligible patients will undergo electrocardiogram based screening for atrial fibrillation, as well as brain natriuretic peptide tests prior to surgery. They will undergo 24 hour holter monitor prior to surgery, and at 30 and 90 days following surgery.

The primary outcome will be occurrence of atrial fibrillation within 90 days of surgery. Secondary outcomes include quality of life change, use of hospital services for atrial fibrillation, and complications of atrial fibrillation. This will be used to validate the pre-existing model for prediction of atrial fibrillation.

DETAILED DESCRIPTION:
Background Atrial fibrillation is an irregularly irregular heartbeat and occurs in around 1.5% of the population. It is associated with negative clinical outcomes such as cardiac failure and mortality. It is strongly implicated in the evolution of stroke, which carries significant burden and cost to patients and the National Health Service (NHS). Atrial fibrillation can be triggered by major physiological stresses such as surgery. The literature suggests that symptomatic atrial fibrillation occurs in 10% of patients within 90 days of surgery. This means that a proportion of patients may have undetected atrial fibrillation, and require treatment to reduce their risk of complications. As the investigators move towards stratified and personalised medicine, it is important to identify the characteristics of the patients at risk of developing atrial fibrillation after surgery in order to mitigate the effects of the condition. This research group has proposed a basic model to stratify patients into high risk groups for post-operative atrial fibrillation, although this requires testing and refinement in a prospective study.

Aims To estimate the rate of atrial fibrillation following colorectal cancer surgery and to characterise patients at highest risk of atrial fibrillation following surgery for colorectal cancer.

Method A prospective study of patients over the age of 65 undergoing colorectal cancer resection will be conducted across 15 colorectal units in the United Kingdom. It will recruit 720 patients over an 18 month period. The study has been designed with regard to public and patient involvement. Patients over the age of 65 undergoing surgery for colorectal cancer with curative intent and no prior diagnosis of atrial fibrillation will be eligible for inclusion. Participants will be screened prior to entry with an electrocardiogram (ECG). Following consent, routine demographic data, EQ-5D-5L (five dimension), and blood sample for Brain Natriuretic Peptide (BNP) will be collected. A 24-hour cardiac rhythm recording will be undertaken prior to surgery to confirm the absences of atrial fibrillation. ECG will be repeated on the day of discharge and 24 hour rhythm recordings repeated at 30 and 90 days post surgery. EQ-5D-5L x will be recorded at 90 days along with any use of health services for cardiac symptoms. Participants diagnosed with atrial fibrillation during the study will be directed to local inpatient or primary care services as appropriate. Demographic characteristics, ECG parameters and BNP will be combined with a previously derived model and tested for ability to predict atrial fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥65 years old
* Undergoing elective surgery for colorectal cancer with curative intent
* No prior diagnosis of atrial fibrillation.
* Willing to consent

Exclusion Criteria:

* Patients aged less than 65 years old
* Pre-existing atrial fibrillation (persistent or paroxysmal)
* Unable to provide informed consent
* Life expectancy <12 months
* Prisoners
* Known pregnancy
* Lack mental capacity
* Patients with limited English language as there is no funding to cover costs of translation of materials

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Colorectal Cancer undergoing elective resection with curative intent.
Sampling Method: Non-Probability Sample
Enrollment: 720 (Estimated)
Dates: Start 2020-01-16 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of atrial fibrillation within 90 days of colorectal cancer surgery, defined as ≥30 seconds of atrial fibrillation identified on a 24-hour cardiac monitor OR absence of p waves and irregularly irregular rhythm on an electrocardiogram | Within 90 days of colorectal cancer surgery
  24-hour recordings will be undertaken at 30 & 90 days post surgery, and electrocardiogram on the day of discharge from hospital.

SECONDARY OUTCOMES:
Quality of life change (EQ-5D-5L (Euroqol-five dimension-five level) | Within 90 days of colorectal cancer surgery
  Quality of life change as measured using EQ-5D-5L from baseline to 90 days post-surgery calculated as population adjusted health index based on total score. In the UK population this can range from -0.594 to 1.0. Higher values are associated with better quality of life scores. A positive change in quality of life index means improved quality of life.
Occurrence of complications of atrial fibrillation | Within 90 days of colorectal cancer surgery
  Includes stroke and embolic events
Number of events of use of health services for atrial fibrillation or sequelae of atrial fibrillation | Within 90 days of colorectal cancer surgery
  Number of events where health services accessed (e.g. primary care, hospital) including for treatment of atrial fibrillation or consequences such as cardiac failure, thromboembolism, or stroke.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Lee, MBChB PhD, Principal Investigator — Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heywood EG, Drake TM, Bradburn M, Lee J, Wilson MJ, Lee MJ. Atrial Fibrillation After Gastrointestinal Surgery: Incidence and Associated Risk Factors. J Surg Res. 2019 Jun;238:23-28. doi: 10.1016/j.jss.2019.01.017. Epub 2019 Feb 5. PMID 30735962
- [Background] Chebbout R, Heywood EG, Drake TM, Wild JRL, Lee J, Wilson M, Lee MJ. A systematic review of the incidence of and risk factors for postoperative atrial fibrillation following general surgery. Anaesthesia. 2018 Apr;73(4):490-498. doi: 10.1111/anae.14118. Epub 2017 Nov 4. PMID 29105078